CLINICAL TRIAL: NCT01471951
Title: Single Human Embryo Transfer: Comparison of Morphologic and Morphometric Parameters for Day 2 Embryo Selection Before Transference.
Brief Title: Single Human Embryo Transfer in Assisted Reproduction Programs
Acronym: SET
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion Para La Investigacion Hospital La Fe (Other)
Responsible Party: Principal Investigator, Inmaculada Molina Botella, Head biologist of the human reproduction unit, Fundacion Para La Investigacion Hospital La Fe
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011/0329
Record Dates: First submitted 2011-11-09; First posted 2011-11-16 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Multiple Pregnancies
MeSH Terms: interventions — Single Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single embryo transfer (Experimental)
  Interventions: Other: Single embryo transfer in women at risk of multiple pregnancies

INTERVENTIONS:
Other: Single embryo transfer in women at risk of multiple pregnancies — Prospective study of single embryo transfers in selected women with good reproductive prognosis and high risk of multiple pregnancies in an IVF-ICSI program.. The day of the embryo transfer, the patients will be randomized by a computer application for morphological and morphometric embryo selection.

SUMMARY:
Embryo selection based on the use of morphometric parameters should increase the implantation success rate.

One of the most important issues of "Assisted Reproduction Technologies (ART)" is the possibility of multiple pregnancies which carries a significant risk for maternal-fetal health. These risks can be reduced by restricting the number of embryos transferred.

To do this, it is essential to improve current techniques of embryo selection by developing new tools that would allow the selection of the embryos with higher implantation potential. In previous works (Molina et al 2011) the investigators have demonstrated greater efficacy for the embryo classification systems based on the use of the morphometric variables. The investigators have also developed a profile of embryo implantation using these morphometric variables. In this project the investigators intend to validate the clinical validity of this new embryo classification system by conducting a prospective study of single embryo transfer (SET) in young women at risk of multiple pregnancies.

ELIGIBILITY:
Inclusion Criteria:

* Personal and family history without interest, not toxic habits.
* Less than 35 years at the time of IVF-ICSI cycle
* Sterility of unknown origin or tubal obstruction.

Exclusion Criteria:

* Repeat nonvoluntary abortions
* Endometriosis
* Polycystic ovary syndrome (criteria Rotterdam 2004)
* Severe male factor (REM <1 million sperm / ml)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 154 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 6 weeks after the embryo transference
  Pregnancy was defined as a gestational sac with a foetus with heart activity detected through sonography in gestational week 6-8.The implantation rate was defined as the number of gestational sacs per number of transferred embryos.

SECONDARY OUTCOMES:
Morphologic embryo selection | 48 hours post insemination (day 2)
  The morphological selection will be made by direct observation of the embryo in an inverted microscope phase contrast. Cell number, blastomere symmetry and fragmentation, and structural abnormalities of the zona pellucida (ZP)were recorded
Morphometric embryo selection | 48 hours post insemination (day 2)
  Morphometric selection will be made by obtaining serial photographs of the embryo that will later be analyzed with an image analysis program that will select the best quality embryos for later transfer The images were analyzed by using ImageJ, a public program developed by Wayne Rasband (http://rsb.info.nih.gov/ij/) and their available tools. The program was used interactively, by applying several of tools and plugins in order to determine the region of interest for the measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Jose J Pertusa, Ph.D., Study Chair — Director of the deparment of Biología Funcional y Análisis de Imagen; Antonio A Pellicer, Ph.D., Study Director — Head of Gynecology and Obstetrics; Inmaculada I Molina, Ph.D., Principal Investigator — Embryologist of the Human Reproduction Unit
Locations (1):
- Hospital Universitari La Fe, Valencia, Valencia, Spain